CLINICAL TRIAL: NCT04578119
Title: Comparison of Sliding Technique and Conventional Technique for Videolaryngoscopy in Patients Undergoing Cervical Spine Surgery With Semi-rigid Neck Collar During Intubation
Brief Title: Optimal Intubating Technique Using Videolaryngoscopy in Patients With Semi-rigid Neck Collar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Do-Hyeong Kim, Associate professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 3-2020-0318
Record Dates: First submitted 2020-09-23; First posted 2020-10-08 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Cervical Spine Surgery; Intubation;Difficult

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Intubating Technique (No Intervention): 'Conventional technique' means that endotracheal intubation is performed with the videolayngoscope blade lifting up the epiglottis.
- Sliding Intubating Technique (Experimental): 'Sliding technique' means that endotracheal intubation is performed by sliding the videolayngoscope blade under the epiglottis smoothly.
  Interventions: Procedure: Sliding Intubating Technique

INTERVENTIONS:
Procedure: Sliding Intubating Technique — Sliding technique' means that endotracheal intubation is performed by sliding the videolayngoscope blade under the epiglottis smoothly.
  Arms: Sliding Intubating Technique

SUMMARY:
In the case of tracheal intubation using a video laryngoscope, both techniques, one is 'conventional technique' in which intubation is performed by placing the blade tip on the vallecula and the other is 'sliding technique' performed by sliding the blade under the epiglottis, are commonly conducted by anesthesiologists. Investigators would like to compare if the sliding technique can improve the condition of tracheal intubation in patients wearing semi-rigid neck collars in cervical spine surgery.

DETAILED DESCRIPTION:
For patients who need to limit the movement of the cervical spine, the tracheal intubation becomes difficult because the head must be positioned in the neutral position. Most of all, with a semi-rigid neck collar that maintains the neutral position of the head and neck, movement is limited and the mouth is not well-opened make the environment of tracheal intubation worse, which result in hypoxia or throat complications related to general anesthesia. Fortunately, it is possible that the development of video laryngoscope assists tracheal intubation easier for patients who have the limited movement of the cervical spine. However, the preferred intubation style and instrument selection for each operator are varied; the established method is required. In the case of tracheal intubation using a video laryngoscope, both techniques, one is 'conventional technique' in which intubation is performed by placing the blade tip on the vallecula and the other is 'sliding technique' performed by sliding the blade under the epiglottis, are commonly conducted by anesthesiologists. Investigators would like to compare if the sliding technique can improve the condition of tracheal intubation in patients wearing semi-rigid neck collars in cervical spine surgery.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients (over 19 years of age) with ASA class I-III undergoing cervical spine surgery at our institution in the department of spine neurosurgery

Exclusion Criteria:

* When rapid sequence induction is required
* When awake intubation is required
* If a subject is on the medication for asthma
* If as subject cannot read or understand the consent form of study

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
percentage of glottic opening (POGO) score (%) | When we insert the endotracheal tube during anesthetic induction
  The POGO score represents the percentage of glottic opening seen, defined by the linear span from the anterior commisure to the interarytenoid notch.

CONTACTS AND LOCATIONS:
Locations (1):
- GangnamSeverance Hospital, Seoul, South Korea